CLINICAL TRIAL: NCT04357236
Title: 18F-FDG PET Imaging Analysis of Antiepileptic Drug Response in Benign Epilepsy With Centrotemporal Spikes Patients
Brief Title: 18F-FDG PET Imaging Analysis of Antiepileptic Drug Response in BECTS
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-437
Record Dates: First submitted 2020-04-20; First posted 2020-04-22 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Benign Epilepsy With Centrotemporal Spikes
Keywords: Benign Epilepsy with Centrotemporal Spikes; glucose metabolism; positron emission tomography; machine learning
MeSH Terms: conditions — Epilepsy, Rolandic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental Group: The experimental group received 18F-FDG PET examination
- Control Group: The control group received 18F-FDG PET examination

SUMMARY:
This original article is a novel investigation on the metabolic characteristics of different patterns of antiepileptic drug (AED) responses in benign epilepsy with centrotemporal spikes (BECTS) patients using 18F-FDG PET imaging. In this study, we demonstrated remitting-relapsing group showed more widespread hypo-metabolism regions than AED responders. Results indicated that metabolic differences had the ability to distinguish the remitting-relapsing patients from AED responders. 18F-FDG PET could be used as a marker to infer the current seizure activity of BECTS. We think that the established hybrid model based on PET and clinical features may be a critical reference for better personalized medication in patients with BECTS.

DETAILED DESCRIPTION:
Purpose The current drug treatment of benign epilepsy with centrotemporal spikes (BECTS) mainly depends on the clinical experience of physicians. This study aimed to investigate different patterns of antiepileptic drug (AED) responses in patients with BECTS using 18F-fluorodeoxyglucose positron emission tomography (18F-FDG PET) imaging for better personalized medication.

Methods A total of 55 patients with BECTS (36 AED responders, 19 remitting-relapsing patients) and 23 pseudo-controls who underwent 18F-FDG PET imaging were retrospectively included. The group comparison was performed to investigate metabolic differences among AED responders, remitting-relapsing patients and pseudo-controls. Three different logistic regression models were employed to distinguish remitting-relapsing patients from AED responders based on clinical features, 18F-FDG PET images and a hybrid of both. Ten AED responders who reduced AED dose and one remitting-relapsing patient who relapsed within one month after PET examination were included in the model evaluation.

ELIGIBILITY:
Inclusion Criteria:

* 1.clinical diagnosis of BECTS; 2. aging between 6 and 18 years ; 3.taking MRI and EEG examination; 4. taking AEDs as prescribed; 5. continuous 12-month clinical follow-up after 18F-FDG PET examination; 6.the last seizure occurring earlier than 24 h before 18F-FDG PET study

Exclusion Criteria:

* 1.any history of neurological disorders, such as head trauma, tumor or infarct

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients with benign epilepsy with centrotemporal spikes
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-04-20 (Actual)

PRIMARY OUTCOMES:
The 'area under curve' (AUC ) of our model in classification performance | Through study completion, about 6 months
  To evaluate the performance of our model, the investigators calculated the AUC of three different logistic regression models based on clinical features, 18F-FDG PET images and a hybrid of both.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nuclear Medicine and PET/CT Center, The Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No